CLINICAL TRIAL: NCT00079118
Title: Phase II Trial of Weekly Irinotecan and Docetaxel in Refractory Metastatic Breast Cancer
Brief Title: Irinotecan and Docetaxel in Treating Patients With Refractory Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0332; NCI-2012-02579 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000354417 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel + irinotecan (Experimental): Patients receive docetaxel IV over 1 hour followed by irinotecan IV over 1 hour on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) receive 2 additional courses beyond CR.
  Patients are followed every 2 months until disease progression and then every 6 months thereafter.
  Interventions: Drug: docetaxel; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: docetaxel
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving irinotecan together with docetaxel works in treating patients with refractory metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of irinotecan and docetaxel, in terms of response rate, in patients with refractory metastatic breast cancer.

Secondary

* Determine the toxicity profile of this regimen in these patients.
* Determine the progression-free and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 1 hour followed by irinotecan IV over 1 hour on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) receive 2 additional courses beyond CR.

Patients are followed every 2 months until disease progression and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Metastatic disease
* Previously treated with chemotherapy in the adjuvant setting and/or for metastatic disease
* At least one unidimensionally measurable lesion

  * At least 20 mm by CT scan or MRI OR at least 10 mm by spiral CT scan
  * Superficial clinical lesions (e.g., skin nodules or palpable lymph nodes) are allowed
  * Lesions on chest x-ray are allowed provided they are clearly defined and surrounded by aerated lung
  * The following are not considered measurable:

    * Bone lesions
    * Ascites
    * Leptomeningeal disease
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Cystic lesions
* No known CNS metastases unless controlled by prior surgery and/or radiotherapy
* Hormone receptor status:

  * Estrogen receptor (ER) and/or progesterone receptor (PR) status known

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Granulocyte count ≥ 1,500/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ upper limit of normal (ULN)
* Meets 1 of the following criteria:

  * AST or ALT ≤ ULN AND alkaline phosphatase ≤ 5 times ULN
  * Alkaline phosphatase ≤ ULN AND AST or ALT ≤ 5 times ULN
  * AST or ALT ≤ 1.5 times ULN AND alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No myocardial infarction within the past 180 days
* No congestive heart failure
* No unstable angina
* No clinically significant pericardial effusion or arrhythmias

Other

* No active, unresolved infection
* No prior severe hypersensitivity reaction to docetaxel, irinotecan, or any drug formulated with polysorbate 80
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No grade 1 or greater sensory or motor neuropathy
* No other concurrent severe condition that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior trastuzumab (Herceptin®) required for HER-2-positive patients (unless contraindicated)

Chemotherapy

* See Disease Characteristics
* More than 14 days since prior chemotherapy
* No more than 2 prior chemotherapy regimens for metastatic disease
* No prior irinotecan or docetaxel for metastatic disease

  * Docetaxel as adjuvant therapy allowed
* No other concurrent chemotherapy

Endocrine therapy

* Prior hormonal therapy required for patients with ER- and/or PR-positive tumors (unless contraindicated)

Radiotherapy

* See Disease Characteristics
* At least 30 days since prior radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* At least 3 weeks since prior major surgery and recovered

Other

* More than 7 days since prior parenteral antibiotic therapy
* No other concurrent experimental drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2004-04; Primary Completion 2007-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Confirmed tumor response as measured by RECIST criteria | Up to 5 years

SECONDARY OUTCOMES:
Distribution of progression times | Up to 5 years
Overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Edith A. Perez, MD, Study Chair — Mayo Clinic
Locations (162):
- United States (162):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Ottumwa Regional Health Center Cancer Center, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - Immanuel St. Joseph's Clinic, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA at Maplewood Cancer Center, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Adult and Pediatric Urology, P.L.L.P., Sartell, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin

REFERENCES:
- [Result] Tan WW, Hillman DW, Salim M, Northfelt DW, Anderson DM, Stella PJ, Niedringhaus R, Bernath AM, Gamini SS, Palmieri F, Perez EA. N0332 phase 2 trial of weekly irinotecan hydrochloride and docetaxel in refractory metastatic breast cancer: a North Central Cancer Treatment Group (NCCTG) Trial. Ann Oncol. 2010 Mar;21(3):493-497. doi: 10.1093/annonc/mdp328. Epub 2009 Jul 22. PMID 19625343